CLINICAL TRIAL: NCT00786344
Title: Health Mediating Effects of the Well Elderly Program
Brief Title: USC Well Elderly Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Florence Clark, PhD, OTR/L, FAOTA; Principal Investigator, USC Division of Occupational Science & Occupational Therapy
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 5R01AG021108-04 (NIH)
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-10

CONDITIONS: Aged
Keywords: Health Promotion: Wellness Programs; Occupational Therapy; Quality of Life; Health; Biomarkers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Redesign (Experimental)
  Interventions: Behavioral: Lifestyle Redesign
- No Treatment Control (No Intervention): The no treatment control arm did not receive the intervention during the first six-month period. However the intervention, which has been proven to be beneficial, was administered to the control arm immediately following the 6 month assessment.

INTERVENTIONS:
Behavioral: Lifestyle Redesign — For a six-month period, each elder participated in weekly 2-hour sessions involving groups of size 8-10, and also received up to 10 hours of individualized treatment over this time period.
  Modular treatment units included the following content areas: (1) Introduction to the Power of Activity; (2) Aging, Health, and Activity; (3) Transportation; (4) Safety; (5) Social Relationships; (6) Cultural Awareness; (7) Finances; and (8) Integrative Summary: Lifestyle Redesign Notebook. The methods of program delivery consisted of didactic presentation, peer exchange, direct experience, and personal exploration. Treatment materials were translated into Spanish and culturally adapted for approximately 15% of the subjects.
  Other Names: Well Elderly Intervention
  Arms: Lifestyle Redesign

SUMMARY:
The purpose of this study is to learn how activity promotes health and well being among older adults. There are two main study goals: (1) to extend the previous results obtained for the Well Elderly Study 1; and (2) to determine what factors make the program successful.

DETAILED DESCRIPTION:
Previous theory and research implicates participation in meaningful activity as an important factor in enhancing older adults' health-related quality of life. Consistent with this emphasis, a previous R01 grant completed by our study group demonstrated that an activity-based intervention (the Well Elderly Intervention) reduced declines in a wide variety of health-related parameters among low income, ethnically diverse elders. In the current four-year project, we attempted to replicate our previous result while simultaneously examining the mediating mechanisms responsible for its positive effects. The outcomes of this study will provide important new information about the process events by which activity-based lifestyle interventions influence key aging outcomes.

In the study, 460 ethnically diverse elders were recruited from 21 sites in the greater Los Angeles area, and participated in a randomized experiment containing a semi-crossover design component. The sites included 9 senior citizen centers (Culver City Senior Center, Estelle Van Meter Multipurpose Center, Hawthorne Senior Center, Hollywood Senior Multipurpose Center, Joslyn Adult Center - Burbank, Lennox Senior Center, Long Beach Senior Center, St. Barnabas Senior Center, and Slauson Recreation Center), as well as 12 senior residences (Casa TELACU, Covenant Manor, Eucalyptus Park, George McDonald Court, Motion Picture and Television Fund, Pilgrim Towers East, Regent Plaza, TELACU Del Rio, TELACU Manor, TELACU Senior Housing, TELACU Terrace, and Ward Villas).

Within either the first or second six-month phase of their study involvement, each subject received a lifestyle-based intervention designed to improve a variety of aging outcomes. At 4-5 points in time over an 18-24 month interval, elders completed assessments of healthy activity, coping, social support, perceived control, stress-related biomarkers, perceived physical health, psychosocial well-being, and cognitive functioning to test the efficacy of the intervention and document the process mechanisms responsible for its effects.

The study has three long-term objectives. First, it will lead to more effective health care services for our nation's rapidly growing elderly population, thereby fulfilling a major policy priority for older adults, namely, preventing declines in their health and independence. Second, it will generate new information regarding how activity influences aging outcomes. Although previous research has shown that activity patterns consistently relate to important aging outcomes, little is known about how the psychological and biological changes that stem from activities combine to promote successful aging. This study will reduce this knowledge gap. Third, due to the significant ethnic diversity at the study sites, the project will produce results that generalize to minority elders. This outcome is important due to the increasing ethnic diversity of our nation's aging population.

ELIGIBILITY:
Inclusion Criteria:

* Fluent speaker of English or Spanish
* Living in the community

Exclusion Criteria:

* Hospitalized
* Living in nursing home
* Mental confusion/dementia
* Participation in the first Well Elderly Study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2004-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Perceived Physical Health | within 1 month of completion of intervention
Psychosocial Well-Being | within 1 month of completion of intervention
Cognitive Functioning | within 1 month of completion of intervention

SECONDARY OUTCOMES:
Healthy Activity | within 1 month of completion of intervention
Active Coping | within 1 month of completion of intervention
Perceived Control | within 1 month of completion of intervention
Social Support | within 1 month of completion of intervention
Positive Reinterpretation-Based Coping | within 1 month of completion of intervention
Stress-Related Biomarkers | within 1 month of completion of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Florence A Clark, PhD, OTR/L, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Leland NE, Fogelberg D, Sleight A, Mallinson T, Vigen C, Blanchard J, Carlson M, Clark F. Napping and Nighttime Sleep: Findings From an Occupation-Based Intervention. Am J Occup Ther. 2016 Jul-Aug;70(4):7004270010p1-7. doi: 10.5014/ajot.2016.017657. PMID 27294991
- [Derived] Clark F, Jackson J, Carlson M, Chou CP, Cherry BJ, Jordan-Marsh M, Knight BG, Mandel D, Blanchard J, Granger DA, Wilcox RR, Lai MY, White B, Hay J, Lam C, Marterella A, Azen SP. Effectiveness of a lifestyle intervention in promoting the well-being of independently living older people: results of the Well Elderly 2 Randomised Controlled Trial. J Epidemiol Community Health. 2012 Sep;66(9):782-90. doi: 10.1136/jech.2009.099754. Epub 2011 Jun 2. PMID 21636614